CLINICAL TRIAL: NCT06008041
Title: Multimodal Epicardial and Endocardial COronary PHYsiological Evaluation in Pathological Situations
Brief Title: Multimodal Epicardial and Endocardial COronary PHYsiological Evaluation in Pathological Situations (PHYCO)
Acronym: PHYCO
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC23.0037 - PHYCO
Record Dates: First submitted 2023-08-16; First posted 2023-08-23 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Coronary Artery Disease; Coronary Microvascular Dysfunction
Keywords: Coronary Artery Disease; Coronary Physiology; Index of Microcirculatory Resistance (IMR)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
When performing coronary angiography in a stable situation, the identification of an intermediate coronary lesion (between 50 and 70%) is common, and requires additional functional evaluation. The gold standard for this evaluation is Fractional Flow Reserve (FFR). FFR is a flow ratio transformed into a pressure ratio by simplification, neglecting some parameters, especially microcirculatory resistance.

The aim of this study is to investigate hemodynamic and structural assessment induced in specific conditions, and their repercussion on functional assessment by FFR to implement the diagnostic approach and personalize it for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate coronary lesion (between 50 and 70%)

Exclusion Criteria:

* Hemodynamic instability
* Adenosine hypersensitivity
* Asthma
* Severe chronic obstructive pulmonary disease
* Long QTc
* Wolff parkinson white
* High degree atriovenricular block
* Left-right shunt
* Carotid artery stenosis with hemodynamic insufficiency
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Diabetes mellitus
  * High blood pressure
  * Aortic stenosis
  * Hypertrophic cardiopathy
  * Dilated cardiopathy
  * Stress cardiopathy
  * Elderly people > 75 years old
  * Acute coronary syndrome
  * Preserved heart failure
  * Cardiac amyloidosis
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Index of Microcirculatory Resistance (IMR) | During coronary angiography
  IMR = Pd x Tmn at maximal hyperhemia Normal range < 25

SECONDARY OUTCOMES:
Fractional Flow Reserve (FFR) | During coronary angiography
  FFR = Pd/Pa at maximal hyperhemia Normal value > 0.80
Coronary Flow Reserve (CFR) | During coronary angiography
  CFR = Hyperhemic flow / Resting flow Normal value > 2
Resting Full cycle Ratio (RFR) | During coronary angiography
  Lowest Pd/Pa value in systole and diastole (mean of 5 consecutive cardiac cycles) Normal value > 0.80
Quantitative Flow Ratio (QFR) | During coronary angiography
  Normal value > 0.80
Angio-IMR | During coronary angiography
  Estimated hyperemic Pa × angio-FFR × [vessel length/(K × Vdiastole)] Normal value < 25
Death | 12 months
Angina pectoris (CCS) | 12 months
  Grade I : Angina with strenuous or rapid or prolonged exertion at work or recreation Grade II : Slight limitation of ordinary activity Grade III : Marked limitation of ordinary physical activity Grade IV : Inability to carry on any physical activity without discomfort, anginal syndrome may be present at rest

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.